CLINICAL TRIAL: NCT00996255
Title: A Phase I Dose-Escalation Study of PHA-793887 Administered as a 1-hour IV Infusion on Days 1, 8 and 15 in a 4-Week Cycle in Patients With Advanced/Metastatic Solid Tumors
Brief Title: Dose-Escalation Study of PHA-793887 in Patients With Advanced/Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Nerviano Medical Sciences (Industry)
Responsible Party: Clinical Research Head, Nerviano Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDKC-887-001; EudraCT Number: 2006-002149-35
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Advanced/Metastatic Solid Tumors
MeSH Terms: interventions — N-(6,6-dimethyl-5-((1-methylpiperidin-4-yl)carbonyl)-1,4,5,6-tetrahydropyrrolo(3,4-c)pyrazol-3-yl)-3-methylbutanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose-Escalation (Experimental)
  Interventions: Drug: PHA-793887

INTERVENTIONS:
Drug: PHA-793887 — Escalating doses of PHA-793887 administered weekly by IV infusion for 3 consecutive weeks in 4-week cycles.

SUMMARY:
The purpose of this open-label, multi center, phase I study, was to determine the safety profile of PHA-793887 administered by intravenous infusion to patients with advanced/metastatic solid tumors. This was a dose-finding study to determine the maximum tolerated dose and the dose of PHA-793887 that can be safely used in phase II investigations.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/metastatic solid tumors for which no standard therapy exists
* ECOG (WHO) performance status 0-1
* Life expectancy of at least 3 months
* Age ≥ 18 years
* Adequate liver, pancreas and renal function
* Acceptable hematologic status
* Acute toxic effects from prior therapy must be resolved to NCI CTCAE Grade ≤ 1
* Treatment with surgery, chemotherapy, or investigational therapy must be completed at least one month prior to treatment initiation (6 weeks for nitrosoureas or Mitomycin C and liposomal doxorubicin)
* Prior radiation therapy allowed in no more than 25% of bone marrow reserve
* Men and women of child-producing potential must agree upon the use of effective contraceptive methods

Exclusion Criteria:

* In the past 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis
* Known brain metastases
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Pregnant or breast feeding women
* Known infection with HIV, active hepatitis B or hepatitis C
* Patients who have exhibited allergic reactions to a similar structural compound, biological agent, or formulation
* History of pancreatitis or disorders making the patient at risk of pancreatitis
* Previous history or current presence of neurological disorders
* Patients with pre-existing symptoms of peripheral neuropathy not related to prior anticancer therapy(ies)
* Concomitant treatment that may be associated with peripheral neuropathy
* Other severe concurrent conditions that could compromise protocol objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Determination of Dose Limiting Toxicities and Maximum Tolerated Dose | First cycle

SECONDARY OUTCOMES:
Assessment of Adverse Events (based on CTCAE version 3.0) | All cycles
Evaluation of pharmacokinetics: plasma concentrations at different times after dosing and related assessment of conventional pharmacokinetic parameters. | First 2 cycles
Evaluation of pharmacodynamics: biomarkers modulation in skin and tumor samples of consenting patients at baseline and post-treatment. | First cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Soria, MD Professor, Principal Investigator — Institut Gustave-Roussy, Villejuif Cedex, France; Chris Twelves, MD Professor, Principal Investigator — St James University Hospital, Leeds, UK
Locations (2):
- Institut Gustave-Roussy, Villejuif, France
- St. James University Hospital, Leeds, United Kingdom